CLINICAL TRIAL: NCT00565149
Title: Dietary Protein Content Determines Weight Gain During High Fat Overfeeding
Brief Title: PROOF: PROtein OverFeeding Effect on Body Weight
Acronym: PROOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Leanne Redman, Professor, Adjunct, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBRC 25007; 2005-34323-15741
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Normal Protein (15%) diet
  Interventions: Behavioral: PROOF
- 2 (Experimental): Low Protein (5%) diet
  Interventions: Behavioral: PROOF
- 3 (Experimental): High Protein (25%) diet
  Interventions: Behavioral: PROOF

INTERVENTIONS:
Behavioral: PROOF — dietary overfeeding with high, low or normal protein content
  Other Names: Overfeeding with different protein levels.

SUMMARY:
This study is designed to determine the effects of dietary protein content on overfeeding.

DETAILED DESCRIPTION:
When body weight increases, the expenditure of energy increases as a mechanism to dissipate the excess calories. The role of diet composition in over-feeding/energy dissipation in humans is unknown. We propose that:

1. High and low protein diet will result in less weight gain as compared to a moderate protein diet during a 56d high fat overfeeding.
2. Increase in energy expenditure and spontaneous physical activity, adjusted for lean and fat mass will be greater in the high and low protein diets as compared to a moderate protein diet.
3. the average size of the fat cells and the pattern of genes expressed in the adipose tissue, skeletal muscle, and peripheral blood mononuclear cells will "predict" which group of subjects will gain the most weight (and fat mass) independent of the level of the protein in the diet.

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI of 19-30kg/m2 A cutpoint of 26kg/m2 will be used to allocate treatment across the three diets. See the statistics section for more detail.
* Are willing to eat all of the study foods even when full
* Are willing to eat only foods provided by Pennington and all of the foods provided
* Are willing to live at Pennington for 10-12 weeks possibly without leaving the metabolic unit the entire time
* Are willing to avoid exercise while in the inpatient phase of the study
* Age 18 - 35

Exclusion Criteria:

Participants are ineligible to participate in the study if they…

* Smoke
* Have Diabetes
* Have claustrophobia
* Have a Fasting Blood Sugar >110
* Have a history of cardiovascular disease
* Have an average screening blood pressure >140/90
* Have a history of a major psychiatric, addictive or eating disorder or any psychosocial or scheduling factors that could impede study outcomes
* Post obese (self-reported BMI) must never have had a BMI greater than 32
* Exercise more than 2 hours per week
* Unable to complete VO2 max test.
* Weight gain or loss of > 3kg in the last 6 months
* Have significant renal, hepatic, endocrine, pulmonary or hematological disease, or a history of gout
* Have had previous GI surgery, Obstructive disease of the GI tract, Hypermotility disorder or a history of problems of impairment of the gag reflex.
* Corticosteroid use in the last 2 Months
* You are pregnant or breastfeeding
* Have Irregular menstrual cycles
* Use Depo-Provera, hormone implant or estrogen replacement therapy
* Have an allergy to PABA (a component of a B-vitamin often found in sunscreen)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2005-03; Primary Completion 2008-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
To determine the effect of overfeeding 40% above energy balance with a low (5%) or high (25%) vs. normal (15%) protein diet on body weight and body composition as well as energy expenditure and its components. | baseline and after 8 weeks of overfeeding

SECONDARY OUTCOMES:
To relate the baseline characteristics of the subjects [fat cell size, pattern of gene expression, body composition, family history of obesity, etc] to the degree of weight / fat gain during overfeeding. | baseline and after 8 Weeks of over feeding

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Smith, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Hochsmann C, Fearnbach N, Dorling JL, Myers CA, Zhang D, Apolzan JW, Stewart TM, Bray GA, Ravussin E, Martin CK. Effect of 8 weeks of supervised overfeeding on eating attitudes and behaviors, eating disorder symptoms, and body image: Results from the PROOF and EAT studies. Eat Behav. 2021 Dec;43:101570. doi: 10.1016/j.eatbeh.2021.101570. Epub 2021 Oct 1. PMID 34655863
- [Derived] Bray GA, Redman LM, de Jonge L, Rood J, Sutton EF, Smith SR. Plasma fatty acyl-carnitines during 8 weeks of overfeeding: relation to diet energy expenditure and body composition: the PROOF study. Metabolism. 2018 Jun;83:1-10. doi: 10.1016/j.metabol.2018.01.019. Epub 2018 Feb 8. PMID 29374510
- [Derived] Bray GA, Redman LM, de Jonge L, Rood J, Sutton EF, Smith SR. Plasma Amino Acids During 8 Weeks of Overfeeding: Relation to Diet Body Composition and Fat Cell Size in the PROOF Study. Obesity (Silver Spring). 2018 Feb;26(2):324-331. doi: 10.1002/oby.22087. Epub 2017 Dec 27. PMID 29280309
- [Derived] Sutton EF, Bray GA, Burton JH, Smith SR, Redman LM. No evidence for metabolic adaptation in thermic effect of food by dietary protein. Obesity (Silver Spring). 2016 Aug;24(8):1639-42. doi: 10.1002/oby.21541. Epub 2016 Jun 29. PMID 27356102
- [Derived] Bray GA, Redman LM, de Jonge L, Rood J, Smith SR. Effect of Three Levels of Dietary Protein on Metabolic Phenotype of Healthy Individuals With 8 Weeks of Overfeeding. J Clin Endocrinol Metab. 2016 Jul;101(7):2836-43. doi: 10.1210/jc.2016-1313. Epub 2016 May 9. PMID 27159194
- [Derived] Bray GA, Redman LM, de Jonge L, Covington J, Rood J, Brock C, Mancuso S, Martin CK, Smith SR. Effect of protein overfeeding on energy expenditure measured in a metabolic chamber. Am J Clin Nutr. 2015 Mar;101(3):496-505. doi: 10.3945/ajcn.114.091769. Epub 2015 Jan 14. PMID 25733634
- [Derived] Gilmore LA, Ravussin E, Bray GA, Han H, Redman LM. An objective estimate of energy intake during weight gain using the intake-balance method. Am J Clin Nutr. 2014 Sep;100(3):806-12. doi: 10.3945/ajcn.114.087122. Epub 2014 Jul 23. PMID 25057153
- [Derived] Lam YY, Redman LM, Smith SR, Bray GA, Greenway FL, Johannsen D, Ravussin E. Determinants of sedentary 24-h energy expenditure: equations for energy prescription and adjustment in a respiratory chamber. Am J Clin Nutr. 2014 Apr;99(4):834-42. doi: 10.3945/ajcn.113.079566. Epub 2014 Feb 5. PMID 24500151
- [Derived] Bray GA, Smith SR, de Jonge L, Xie H, Rood J, Martin CK, Most M, Brock C, Mancuso S, Redman LM. Effect of dietary protein content on weight gain, energy expenditure, and body composition during overeating: a randomized controlled trial. JAMA. 2012 Jan 4;307(1):47-55. doi: 10.1001/jama.2011.1918. PMID 22215165